CLINICAL TRIAL: NCT06941103
Title: Effects of Spinal Stabilization Exercise Training in Women With Chronic Constipation
Brief Title: Spinal Stabilization Exercise Training in Women With Chronic Constipation
Acronym: Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Özel Artı Disleksi Özel Eğitim ve Rehabilitasyon Merkezi (Other)
Responsible Party: Principal Investigator, Saliha Beste BÜLBÜL, Ankara Yildirim Beyazit University, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Spinal Stabilization Exercise
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Constipation
Keywords: spinal stabilization exercise; quality of life; spinal stability
MeSH Terms: conditions — Constipation | interventions — Health Planning Guidelines

STUDY DESIGN:
Intervention Model Description: Two groups with a control group (recommendation) and exercise group (recommendation+Spinal stabilization exercise training)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Spinal stabilization exercise training group will receive exercise sessions and outcome assessments will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Spinal stabilization exercise training and recommendation
  Interventions: Other: Spinal stabilization exercise training and recommendation; Other: Recommendation
- Control group (Other): Recommendation
  Interventions: Other: Recommendation

INTERVENTIONS:
Other: Spinal stabilization exercise training and recommendation — Spinal stabilization exercise training will be applied 3 days a week for 8 weeks under the supervision of a specialist physiotherapist. Exercises consist of a 5-10 minute warm-up period, 40 minutes SSET and a 5-10 minute cool-down period.
  Within the scope of the recommendation, information will be given about the definition of constipation, risk factors, and treatment methods.. A brochure will be prepared to be distributed to individuals regarding these issues.
  Arms: Exercise group
Other: Recommendation — Within the scope of the recommendation, information will be given about the definition of constipation, risk factors, and treatment methods.. A brochure will be prepared to be distributed to individuals regarding these issues.

SUMMARY:
This study was planned to investigate the effects of spinal stabilization exercise training on constipation symptom severity, quality of life, perception of recovery, and spinal stability in women with chronic constipation.

DETAILED DESCRIPTION:
This study was planned to investigate the effects of spinal stabilization exercise training on constipation symptom severity, quality of life, perception of recovery and spinal stability in women with chronic constipation. Individuals' physical, demographic, lifestyle, medical characteristics and medications used will be questioned and recorded. Physical activity level will be questioned with the "International Physical Activity Questionnaire-Short Form (IPAQ-SF)". In addition, constipation severity will be evaluated before and after treatment with the "Constipation Severity Scale (CSS)", functional markers of the intestine "Stool Diary and Bristol Stool Scale", the effect of constipation on the quality of life "The Patient Assessment of Constipation Quality of Life (PAC-QOL)", spinal stability "Sahrmann Test" and trunk muscle endurance "McGill Core Endurance Tests". In addition, perception of recovery will be evaluated after treatment with the "Patient Global Impression of Improvement Scale" and compliance with the recommendation will be evaluated with the "Visual Analog Scale (VAS)". The control group will be given only suggestions, while the exercise group will be given suggestions and spinal stabilization exercise training. Within the scope of the recommendation, you will first be informed about the definition of constipation, risk factors, treatment methods, and recommendations on physical activity, nutrition (fiber and fluid intake) and defecation position will be given to reduce constipation complaints. A brochure will be prepared to be distributed to individuals regarding these issues. Spinal stabilization exercise training will be applied 3 days a week for 8 weeks under the supervision of a specialist physiotherapist. Exercises consist of a 5-10 minute warm-up period, 40 minutes spinal stabilization exercise training a 5-10 minute cool-down period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic functional constipation according to Rome 4 diagnostic criteria
* Those between the ages of 18-65
* Women who volunteer to participate in the study will be included.

Exclusion Criteria:

* Those who are pregnant or breastfeeding
* Neurological diseases (Parkinson, Multiple Sclerosis, hemiplegia, etc.)
* Undercontrolled systemic/metabolic diseases (hypothyroidism, diabetes mellitus, hypokalemia, hypercalcemia, hypomagnesemia, etc.)
* Malignant diseases
* Accompanying colon or gastrointestinal problems (gastrointestinal bleeding, acute inflammation, etc.)
* Secondary constipation presence of alarm symptoms (new onset constipation, rectal bleeding, involuntary weight loss, nausea, vomiting, fever, anemia or a family history of gastrointestinal malignancy)
* Those who received treatment (exercise, surgery, etc.) for the abdominolumbopelvic region in the last year
* Having a history of colostomy or colectomy
* Those with orthopedic limitations that would affect spinal stabilization exercise training
* Those who do not participate in the treatment program regularly.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Constipation Severity Scale (CSI) | two weeks
  Scale Varma et al. it was developed by to determine individuals' defecation frequency, intensity and difficulty experienced during defecation. Kaya et al. Turkish validity and reliability were conducted by . The scale consists of 16 questions and three sub-areas. These areas are 1. Fecal Obstruction, 2. Large Intestinal Laziness and 3. Pain. The lowest total score that can be obtained from the scale is 0 and the highest is 73. A high score indicates that the symptoms are serious.

SECONDARY OUTCOMES:
Spinal Stability Assessment | two weeks
  Spinal stability will be evaluated with the Sahrmann test and McGill trunk muscle endurance tests.
  In the Sahrmann test, the Stabilizer Pressure Biofeedback Unit (Chattanooga, TN, USA) will be placed under the individuals' lumbar region and adjusted to 40mmHg. Individuals will be taught the abdominal bracing maneuver to ensure isolated contraction of the transversus abdominis muscle and spinal stability. Individuals will be asked to maintain abdominal bracing and perform different lower extremity movements at all levels of the test. The test consists of 5 levels and the difficulty level increases from level 1 to level 5. When the stabilizer value deviates more than 10 mmHg at each level, the test will be terminated, assuming that the person cannot complete that level.In McGill trunk muscle endurance tests, individuals will be subjected to trunk flexion, extension, right and left lateral flexion endurance tests.
Patient Assessment Constipation-Quality of Life Scale (PAC-QOL) | two weeks
  Marquis et al. it was developed by (Marquis et al., 2005) in 2005, and its Turkish validity and reliability were tested by Dedeli et al. It was revealed by. The scale consists of 28 items and has 4 subdomains: "physical discomfort", "psychosocial discomfort", "worry/anxiety" and "satisfaction". The lowest score that can be obtained from the scale is 28 and the highest score is 140. Higher scores from the scale mean that the quality of life is more negatively affected.
Bowel diary | two weeks
  Individuals will be asked to complete a bowel diary one week before starting treatment and for 7 days after the study is completed. In these diaries, they will be asked to mark each day they defecate, how long they spend in the toilet for each defecation, the feeling of incomplete defecation, the use of medication to defecate, changes in nutrition and fluid consumption, and pain during defecation . They will also be asked to record stool type according to the Bristol Stool Scale in their bowel diary. This scale was developed by Lewis and Heaton and human feces are classified into 7 groups. Since the shape of the stool changes depending on the time it stays in the colon, it is a rapid and reliable indicator of colonic transit time. Stool type will be determined according to the data obtained from the scale.
Patient Global Impression of Improvement Scale | two weeks
  Individuals' perception of improvement in constipation complaints at the end of treatment will be questioned with the "Patient Global Impression of Improvement Scale" as follows. "How would you describe your current condition in terms of constipation compared to your condition at the beginning of treatment?" The available answers to this question are "Much better (1)", "Better (2)", "Somewhat better (3)", "No change (4)", "Somewhat worse (5)", "Worse (6)" and "Much worse (7)". Individuals will be asked to mark the answer that best describes their condition among the available answers.
Visual Analog Scale (VAS) | two weeks
  After the treatment, the physical activity, nutrition (fiber and fluid intake) recommendations and compliance with the recommendations given regarding defecation position will be evaluated with the "Visual Analog Scale (VAS)". Individuals will be asked to mark the point that best describes them on a horizontal line with a real length of 10 cm. The distance of the marked point to the "0" point will be measured with a ruler and recorded in cm. On this scale, the "0" point will be defined as "I did not comply at all (%0)" and the "10" point will be defined as "I showed complete compliance (%100)".

CONTACTS AND LOCATIONS:
Locations (1):
- Özel Artı Disleksi Özel Eğitim ve Rehabilitasyon Merkezi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No